CLINICAL TRIAL: NCT04390490
Title: Clinical Trails of Photoelectrochemical Immunosensor for Early Diagnosis of Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bin He (Other)
Responsible Party: Sponsor-Investigator, Bin He, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: XH-20-007
Record Dates: First submitted 2020-05-09; First posted 2020-05-15 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Automatic chemiluminescence analyzer will be used for dectecting the concentration of cardiac troponin I as control group.
- Photoelectrochemical immunosensor (Experimental): Photoelectrochemical immunosensor will be used for dectecting the concentration of cardiac troponin I as test group.
  Interventions: Device: Graphene quantum dots combined with Si nanowire photoelectrochemical immunosensor

INTERVENTIONS:
Device: Graphene quantum dots combined with Si nanowire photoelectrochemical immunosensor — Graphene quantum dots combined with Si nanowire is a new method of photoelectrochemical immunosensor
  Arms: Photoelectrochemical immunosensor

SUMMARY:
The aim of this prospective randomized controlled clinical trial will evaluate the sensitivity, precision and effectiveness of photoelectrochemical immunosensor for early diagosis of acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Symptoms of chest pain

Exclusion Criteria:

* Patients who will undergo immediate PCI Pregnant
* Lactating women
* Patients with mental disorders
* Patients are using other experimental drugs; Refusal to provide informed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of photoelectrochemical immunosensor | 28 days
  Sensitivity，precision and cost of the photoeletrochemical immunosensor

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China